CLINICAL TRIAL: NCT05290272
Title: Validity of AI in Treatment of the Musculoskeletal Conditions by Vifive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: ViFIVE Inc. (Unknown)
Responsible Party: Principal Investigator, Eugene Roh, Clinical Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63794
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Shoulder Adhesive Capsulitis; Knee Osteoarthritis
MeSH Terms: conditions — Bursitis; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ViFIVE Digital Care Program (Experimental): AI based digital care program that is individually tailored for each user depending on need. ViFive DCP includes illustration, voice guidance, and pose correction features of AI coach. Participants will required to complete the program.
  Interventions: Device: ViFIVE Digital Care Progrma

INTERVENTIONS:
Device: ViFIVE Digital Care Progrma — ViFive DCP (Digital Care Program) is a highly structured, protocolized, and individually tailored intervention consisting of personalized exercise therapy modules. ViFive DCP is delivered by a physical therapy team consisting of DPTs and a personal coach. The DCP consists of ten modules and its advancement will be determined by each patient's progress after the treatment team's review every week.
  Other Names: ViFIVE DCP

SUMMARY:
The purpose of this study is to evaluate the efficacy of the 12-week ViFive program, a vision-based artificial intelligent digital care plan for chronic knee pain. ViFive digital care plan is delivered by a physical therapy team consisting of physical therapists and a personal coach. We aim to understand the safety and efficacy of this vision artificial intelligent based home exercise program.

DETAILED DESCRIPTION:
This study is recruiting patients who present with knee osteoarthritis and shoulder adhesive capsulitis through evaluation by the treating physician. A brief physical functional assessment will be conducted to ensure eligibility and assess for any safety concerns (e.g., minimum strength and capability to conduct basic rehabilitation exercises).

Once subject is enrolled and device is distributed and set up, participants will follow and complete the VIFive program on the device.

ViFive DCP (Digital Care Program) is a highly structured, protocolized, and individually tailored intervention consisting of personalized exercise therapy modules. ViFive DCP is delivered by a physical therapy team consisting of DPTs and a personal coach. The DCP consists of ten modules and its advancement will be determined by each patient's progress after the treatment team's review every week. The primary aim of ViFive DCP is to assist patients in recovering their appropriate daily physical activity level by strengthening the knee and educating proper interpretation of sensation rather than pain. ViFive DCP represents a mobile intervention platform utilizing vision-AI. Vision AI enables objective and precise exercise prescription along with transparent patient monitoring. As a platform, there is an interface for patients and clinicians. Each module consists of a specific exercise treatment plan, educational articles, and instructions to promote changes in daily life. Each of these modules has specific goals, and patients are able to follow a predefined sequence of modules. ViFive DCP includes illustration, voice guidance, and pose correction features of AI coach. During treatment, patients have regular contact with their personal coach through a message functioning (e.g., exercise progress, answers to questions, patient receives feedback from the coach, can ask the coach questions, etc). The coach provides continuous feedback on completed tasks and responds to concerns the patient may have. Weekly feedback on progress is also provided. In total, the coach spends approximately 12 hours per patient throughout treatment.

After completion of the program, device will be returned.

Participants are to complete questionnaires, consisting of KOOS, VAS, and surgery interest at baseline, 3-month, and 6-month. VAS will be used to assess changes in pain level. KOOS will be used to assess knee functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 18-60 years old
* Diagnosis of adhesive capsulitis or
* Diagnosis of knee osteoarthritis

Exclusion Criteria:

* Age <18 or >60 years old
* acute injuries or recent surgeries to the knee or shoulder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Score | 6 months
  Patient reported outcome measure that reports a normalized score (100 indicating no symptoms and 0 indicating extreme symptoms). 100 indicating the best score, and 0 indicating the worst score.
Visual Analogue Scale | 6 months
  Patient reported outcome measure that reports pain intensity on a scale of 0-10 (10 being extreme pain and 0 no pain at all). 10 indicating the worst score and 0 indicating the best score.

SECONDARY OUTCOMES:
Surgery Interest | 6 months
  Patient reported outcome measure determining participant's interest in surgery on a scale of 1 to 10 (10 being very interested and 1 being not at all interested).

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Hospitals and Clinics, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: Undecided